CLINICAL TRIAL: NCT07033923
Title: Neuro-computational Study of Thymic Fluctuations in Mood Disorders - MOODELING
Brief Title: Neuro-computational Study of Thymic Fluctuations in Mood Disorders
Acronym: MOODELING
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier St Anne (Other)
Collaborators: Institut du Cerveau et de la Moelle (ICM Institute) (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: D23-P014
Record Dates: First submitted 2025-02-26; First posted 2025-06-24 (Actual); Last update posted 2025-06-24 (Actual); Status verified 2025-06

CONDITIONS: Depression; Bipolar Disorder; Recurrent Depression; Mood Disorders
Keywords: cognitive neuroscience; patient-specific modelling; psychiatry; mood disorders; affective disorders; computational modelling; computational psychiatry; prognosis; predictive medicine
MeSH Terms: conditions — Depression; Bipolar Disorder; Mood Disorders | interventions — Magnetic Resonance Imaging

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- BD Group: patients with bipolar disorder (Experimental): Patients with:
  * a diagnosis of bipolar mood disorder (F31) according to ICD-10 criteria, made by a psychiatrist
  * a thymic episode (F31.0 - F31.6) diagnosed in the past 12 months by a psychiatrist
  Interventions: Diagnostic Test: Brain magnetic resonance imaging (MRI) with structural (anatomical) and functional sequences (optional); Behavioral: Computerized cognitive tests; Device: Daily longitudinal monitoring by mobile MOODELING application

INTERVENTIONS:
Diagnostic Test: Brain magnetic resonance imaging (MRI) with structural (anatomical) and functional sequences (optional) — Brain MRI with structural (anatomical) and functional sequences (without contrast injection) will be collected. The cognitive tests will be carried out during the recording of the functional MRI (optional) in order to highlight the neural correlates of mood variations.
Behavioral: Computerized cognitive tests — Cognitive tests can be administered during the recording of a functional MRI, in order to highlight the neural correlates of mood variations.
  Cognitive data from a computerized experimental psychology experiment: this test involves different tests on a computer or tablet, including a test evaluating the minimal variations in the subject's mood and motivational state during the task, as well as its decision-making abilities.
Device: Daily longitudinal monitoring by mobile MOODELING application — Daily longitudinal monitoring by mobile MOODELING application (mood, energy, events) with self-monitoring tools (calendar, mood curve) at home. Follow-up duration on the application: 12 months

SUMMARY:
Depression and bipolar disorder are frequent, debilitating conditions. Both are thought to be primarily caused by an impaired regulation of mood, which is why they are sometimes referred to as "mood disorders". However, the biological basis of mood remains poorly understood, which is a major limitation for the development of new treatments.

Recent work that combines neuroscience with mathematical models are promising to better understand mood and to link it to its biological basis, but they don't have any medical application yet. Can these models describe mood in a way that is relevant to mood disorders, and help doctors and psychologists predict subsequent clinical evolution? With the objective of extending this framework to real-life fluctuations and to assess its clinical relevance, this study will combine a neuroimaging session with a smartphone-based, longitudinal follow-up. Three groups of 96 subjects each will be recruited: depressive disorder, bipolar disorder and healthy controls. They will have their mood fluctuations assessed first in the lab (in the neuroimaging experiment), then in their daily lives (by providing a few ratings and choices every day on the smartphone app).

This study will allow to better understand the differences in how patients' mood reacts to daily events, as compared to people who don't suffer from depression or bipolar disorder. The combination of the two steps will allow to assess whether a short neuroimaging evaluation can be useful to predict subsequent clinical evolution during the following months.

The investigators wanted to add two optional ancillary studies. The first uses a mobile application for implicit, passive, and longitudinal mood assessments through emotion tracking. Indeed, it seems relevant to add this type of evaluation alongside explicit assessments to more accurately detect mood fluctuations.

The second study uses a mobile application that allows voice recordings. The analysis of these vocal parameters will help to characterize a specific linguistic and vocal profile within the three groups, as well as to identify specific symptoms of conditions such as depression and bipolar disorder.

These ancillary studies will be offered to both patients and the control group.

DETAILED DESCRIPTION:
Mood disorders are common diseases that represent the first psychiatric cause of morbidity and mortality, and a major public health and medico-economic issue at the national and international level.

Although effective treatments exist, understanding of the pathophysiology of these diseases remains largely incomplete. The assessment is entirely clinical, without any reliable biological marker which has serious consequences in terms of morbidity.

Neurocomputational approaches, which consist of describing the cognitive mechanisms underlying the symptoms on which the clinic is based, so as to better articulate them with their biological substrates, are proving promising in the field.

The first mood models mathematically describe the intuitive idea that positive events have a positive impact on mood, and vice versa for negative events. More recent work has developed models to characterize the interaction of mood with decision-making. They describe how mood affects the perception of events and influences the resulting decisions: when mood is high, subjects tend to overestimate potential gains and underestimate losses, and vice versa when mood is low.

The investigators recently replicated these results and identified the neural bases of this phenomenon by showing, using a functional MRI (fMRI) study in healthy volunteers, that mood was encoded in the activity of two brain regions, the ventromedial prefrontal cortex (vmPFC) and the anterior insula (aIns). The activity of these regions in turn modulated the participants attitude towards risky choices. The investigators recently replicated this result in an intracerebral stereo-electroencephalogram (sEEG) study.

The neurocomputational approach to mood has therefore already made it possible:

1. to clarify the reciprocal interactions between mood and decision-making and
2. to propose a first characterization of the neural bases of mood.

This double advance constitutes a first step towards a true mechanistic explanation of mood disorders.

However, these models validated in the context of experiments carried out in the laboratory on healthy volunteers suffer from two limitations. They were used (1) on a short time scale (one hour) compared to daily fluctuations which evolve over a few days or weeks (2) to account for minimal, barely perceptible fluctuations, while the fluctuations observed in the context of mood disorders are extremely intense. To demonstrate their clinical relevance, it is necessary to make a double change of scale, in terms of time and amplitude.

With the aim of bridging this explanatory gap, this study aims to make this change in scale, by including patients and using a mobile application to conduct long follow-up (12 months). Indeed, the use of mobile applications has emerged in recent years as a promising approach, used in several studies with encouraging results, to collect data in ecological conditions (longitudinal, multidimensional monitoring, large samples).

To this end, the investigators will recruit 588 subjects, in 4 groups :

* 96 patients with depressive disorder (DD)
* 96 patients with bipolar disorder (BD)
* 96 healthy controls, as a reference group for comparison
* 300 non selected subjects from the general population.

After receiving written and oral information on the research, how it will be carried out and what their participation will entail, participants can be enrolled in the protocol if they have no exclusion criteria.

At inclusion, socio-demographic, clinical and therapeutic data will be collected, and updated at each visit.

An initial visit with a cognitive assessment will be carried out for patients and controls. For those who accept it, and in whom MRI is not contraindicated, this assessment will be performed during a functional MRI of the brain.

Minimal mood fluctuations will be measured using the feedbacks of a reasoning task, and a decision-making task will be used to reveal their effects on decision-making. Subjective mood ratings provided during this (short-term) lab-experiment will be fitted with our computational model of mood. The investigators will thus obtain, for each participant, a computational fingerprint describing how positive and negative events are integrated into a mood signal. Thus, a first step will be to investigate to what extent this computational fingerprint of mood differs between groups of patients, and compared to healthy controls.

All patients and healthy subjects will then be monitored daily for one year, via a dedicated mobile application. All participants will be required to complete a 3-minutes evaluation on a daily basis. The investigators will collect three types of longitudinal data: subjective mood ratings, positive and negative life events (valence and intensity of the most salient event of the day) and economic choices involving sensitivity to reward, loss, risk, delay, and effort (e.g. do the participant prefers 10 euros now or 20 euros in one week?). As in short-term data, the investigators will obtain, for each participant, a computational fingerprint describing how of positive and negative event are integrated into a mood signal. The investigators predict to observe the same group differences than in short term data: a higher reciprocal effect of mood on the perception of life events in patients with bipolar disorder, and a higher asymmetry between positive and negative life events in patients with recurrent depressive disorder.

Though informative in themselves about the effect of syndromic or sub-syndromic mood fluctuations on decision-making, the investigators also aim to use this ambulatory tool to anticipate relapses in these stabilized patients. Given the frequency of mood relapse in these patients and based on our preliminary data, the investigators expect to observe an actual episode in around one third of them during this 12-month follow-up. Importantly, referring psychiatrists will not have access to the collected data during this follow-up (no risk to alter the usual care), allowing us to test to what extent any of our measures is sensitive and specific enough to predict relapses. A trivial prediction is a shift in mood rating will be observed a few days before actual relapse. However, recent results suggested that decision-making tests could be more sensitive than auto or hetero-questionnaires to detect relapse.

Intermediate visits will be carried out every 3 months, with repeated clinical scales. An end-of-study visit will take place 12 months after inclusion.

The combination of these two steps, first a lab-recorded experiment, then a 12-month follow-up, is a key aspect of this study. Critically, the investigators will compare the computational phenotypes obtained in the very same patients but fitting short-term (a few dozens of minutes) or long-term (12 months) subjective mood ratings. The investigators will investigate to what extent the computational phenotype obtained during the short-term evaluation (first step) is informative about subsequent clinical (and subsyndromic) mood fluctuations.

Finally, a group of healthy volunteers will be monitored only online via the mobile application. This group will allow us to show the validity and stability of computational phenotypes of mood and decision-making, and to calibrate population-based measures of these relevant measures.

In addition, the investigators wanted to add two optional ancillary studies. The first uses a mobile application for implicit, passive, and longitudinal mood assessments through emotion tracking. Indeed, it seems relevant to add this type of evaluation alongside explicit assessments to more accurately detect mood fluctuations.

The second study uses a mobile application that allows voice recordings. The analysis of these vocal parameters will help to characterize a specific linguistic and vocal profile within the three groups, as well as to identify specific symptoms of conditions such as depression and bipolar disorder.

These ancillary studies will be offered to both patients and the control group.

ELIGIBILITY:
Inclusion Criteria:

Common between groups (DD, BD, control and GP):

* Having given informed and written consent
* Being covered by social security

For patients with depressive disorder (DD):

* Having been diagnosed with characterized depressive episode (F32, F33, F34) according to the ICD-10, by a psychiatrist, or having presented this diagnosis during the past 12 months

For patients with bipolar disorder (BD):

* Presenting a diagnosis of bipolar mood disorder (F31) according to ICD-10, by a psychiatrist
* Having presented a mood episode (F31.0 - F31.6) diagnosed during the past 12 months by a psychiatrist

Exclusion Criteria:

Common between groups (DD, BD, control and GP):

* Inability to carry out daily monitoring on mobile application for 12 months
* legal protection measure (guardianship or curatorship)

For control group:

* Current diagnosis of psychiatric disorder in ICD-10 (F20-F98) or prescription of psychotropic treatment
* History of depression (F32)
* Syndrome of dependence on a psychoactive substance other than tobacco
* Neurological history (in particular history of stroke, coma, epilepsy, neuro- inflammatory, or neuro-degenerative disease)
* Inability to carry out daily monitoring on mobile application for 12 months

For patients and healthy volunteers for whom an MRI (without injection of contrast agent) is proposed

* Contraindication to MRI: cardiac pacemaker not compatible with MRI, heart valve implant, implant or metallic foreign body
* Pregnant woman (at the time of MRI)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 588 (Estimated)
Dates: Start 2024-07-18 (Actual); Primary Completion 2028-07-18 (Estimated); Study Completion 2029-07-18 (Estimated)

PRIMARY OUTCOMES:
Computational phenotypes of daily mood fluctuations in the 3 groups | From enrolment to Month 12
  Computational phenotypes of daily mood fluctuations obtained from daily collection of mood data and daily life events via the mobile application.

SECONDARY OUTCOMES:
Short-term computational phenotypes of mood | Month 0
  Computational phenotypes obtained from the mood signal recorded on a short-term assessment (1 hour) measured at inclusion (Month 0) from a cognitive task
Correlation of computational phenotypes of mood at short and long-term | From enrollment to Month 12
  Correlation between computational phenotypes of mood signal obtained from the collection of mood data and daily life events via the mobile application:
  * at short-term (Month 0 - Inclusion)
  * at long-term (Month 12), tested at individual level within each group (DD, BD and control).
Basal fMRI signal characteristics of the vmPFC and aIns in each group | Month 0
  fMRI signal characteristics (BOLD) in the ventromedial prefrontal cortex (vmPFC) and anterior insula (aIns)
Neural correlates from functional MRI (fMRI) | Month 0
  fMRI signal BOLD
Effect of mood on decision-making at short and long-term | From enrolment to Month 12
  Decision-making will be assessed from data collected daily in the mobile application Mood fluctuations will be assessed from data collected daily in the mobile application
Sensitivity of decision-making parameters to predict clinical relapses | Month 0, Month 3, Month 6, Month 9, Month 12
  Clinical relapses assessed by clinical interview
Number of hour per day of sunshine | From enrolment to Month 12
  Daily sushine duration calculated from weather data based on the geographic area of the participant

CONTACTS AND LOCATIONS:
Overall Officials: Fabien Vinckier, Dr, Principal Investigator — GHU Paris Psychiatry & Neurosciences
Locations (2):
- France (2):
  - - Groupe hospitalo-universitaire Paris Psychiatrie et Neurosciences, Paris, Paris
  - Assistance Publique - Hôpitaux de Paris GH Pitié-Salpêtrière, Paris

IPD SHARING:
Plan to Share IPD: Yes
The data obtained from medical visits (clinical informations, biological assessments, cognitive data) and brain MRIs will be kept, coded and archived for a period of two years after the last publication of the research results or until the final research report is signed. These can be used later for collaborative research (academic and/or industrial partners) in the European Union (EU) and/or abroad exclusively for scientific purposes.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: The data obtained from medical visits (clinical informations, biological assessments, neurocognitive data)and brain MRIs will be kept, coded and archived for a period of two years after the last publication of the research results or until the final research report is signed.
Access Criteria: The data can be used for collaborative research (academic and/or industrial partners) in the European Union (EU) and/or abroad exclusively for scientific purposes. Any party must contact the sponsor, who has full property of the data.
  In case of requested transfer of the anonymized database resulting from this research abroad (outside the EU), the sponsor will request information regarding data storage and management, to make sure that the other party will be able to ensure a level of security equivalent to French or European Union law.

REFERENCES:
- [Background] Rutledge RB, Moutoussis M, Smittenaar P, Zeidman P, Taylor T, Hrynkiewicz L, Lam J, Skandali N, Siegel JZ, Ousdal OT, Prabhu G, Dayan P, Fonagy P, Dolan RJ. Association of Neural and Emotional Impacts of Reward Prediction Errors With Major Depression. JAMA Psychiatry. 2017 Aug 1;74(8):790-797. doi: 10.1001/jamapsychiatry.2017.1713. PMID 28678984
- [Background] Eldar E, Rutledge RB, Dolan RJ, Niv Y. Mood as Representation of Momentum. Trends Cogn Sci. 2016 Jan;20(1):15-24. doi: 10.1016/j.tics.2015.07.010. Epub 2015 Nov 3. PMID 26545853
- [Background] Eldar E, Niv Y. Interaction between emotional state and learning underlies mood instability. Nat Commun. 2015 Jan 21;6:6149. doi: 10.1038/ncomms7149. PMID 25608088
- [Background] Heerema R, Carrillo P, Daunizeau J, Vinckier F, Pessiglione M. Mood fluctuations shift cost-benefit tradeoffs in economic decisions. Sci Rep. 2023 Oct 24;13(1):18173. doi: 10.1038/s41598-023-45217-w. PMID 37875525
- [Background] Pessiglione M, Heerema R, Daunizeau J, Vinckier F. Origins and consequences of mood flexibility: a computational perspective. Neurosci Biobehav Rev. 2023 Apr;147:105084. doi: 10.1016/j.neubiorev.2023.105084. Epub 2023 Feb 9. PMID 36764635
- [Background] Vinckier F, Rigoux L, Oudiette D, Pessiglione M. Neuro-computational account of how mood fluctuations arise and affect decision making. Nat Commun. 2018 Apr 26;9(1):1708. doi: 10.1038/s41467-018-03774-z. PMID 29700303
- [Background] Rutledge RB, Skandali N, Dayan P, Dolan RJ. A computational and neural model of momentary subjective well-being. Proc Natl Acad Sci U S A. 2014 Aug 19;111(33):12252-7. doi: 10.1073/pnas.1407535111. Epub 2014 Aug 4. PMID 25092308
- See also: Website of the Moodeling smartphone application used in the study — https://moodeling.icm-institute.org/